CLINICAL TRIAL: NCT05946811
Title: The Role of MACitentan on the Prevention of Residual Pulmonary vasculaR Occlusion
Brief Title: Macitentan to Prevent PRVO
Acronym: MAC-PRO
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was cancelled by funding agency before starting enrollment.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Rafael Cires-Drouet, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00106867
Record Dates: First submitted 2023-06-26; First posted 2023-07-14 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Embolism
Keywords: macitentan; pulmonary embolism; pulmonary hypertension; post-PE syndrome
MeSH Terms: conditions — Pulmonary Embolism; Hypertension, Pulmonary | interventions — macitentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Macitentan arm (Experimental): Participants allocated to this arm will receive Macitentan 10 mg daily for 3 months
  Interventions: Drug: Macitentan 10mg
- Placebo (Placebo Comparator): Participants allocated to this arm will receive placebo daily for 3 months.
  Interventions: Drug: Macitentan 10mg

INTERVENTIONS:
Drug: Macitentan 10mg — Macitentan 10 mg oral once daily for 3 months. vs placebo

SUMMARY:
About half of patients who suffer of a pulmonary embolism (blood clots in the lungs), do not clear completely the clots overtime, increasing the risk of having a new blood clot in the lungs and elevated blood pressure in the pulmonary artery; therefore, developing fatigue, shortness of breath, and heart failure.

The objective of this clinical trial is to compare 3 months of daily Macitentan (a medicine to increase the diameter of the pulmonary artery) in addition to blood thinners vs. blood thinners alone in patients with acute blood clots in the pulmonary artery:

Question 1: Whether the use of Macitentan in addition to blood thinners enhances the process of cleaning the blood clot in the pulmonary artery compared to blood thinners alone.

Question 2: Whether the use of Macitentan in addition to blood thinners is associated to improve the fatigue and shortness of breath in patients after a pulmonary embolism compared to blood thinners alone.

Participants will be asked to take a capsule for 3 months in addition to blood thinners. The capsule could contain either Macitentan (medicine) or a placebo (not medicine). In 3 months, participants will have a new image of the pulmonary artery to document the cleaning of the clots. Also, blood and urine samples will be collected, as well as a questionnaire will be filled out. In 6 months, patients will have repeated images of the heart as well as repeated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old.
* Acute high-risk or intermediate-risk PE diagnosed by CTPA within 28 days prior to enrollment

Exclusion Criteria:

* Contraindication for anticoagulation
* Allergy or contraindications to Macitentan or any other endothelin receptor antagonist.
* Surgical interventions to treat PE including catheter-directed thrombolysis, catheter-based thrombectomy, or surgical pulmonary embolectomy.
* Known inherited or acquired hypercoagulable states
* History of pulmonary embolism prior to index PE
* History of pulmonary hypertension including Group 1 (Primary pulmonary hypertension), Group 2 (secondary to left heart disease), Group 3 (secondary to lung disease), Group 4 (Chronic thromboembolic pulmonary hypertension)
* Severe chronic obstructive pulmonary disease
* Severe uncontrolled asthma
* Pregnancy or fertility treatment
* Breastfeeding
* Life expectancy is less than 6 months
* History of radiation therapy to the chest
* Current or previous use within 90 days of an endothelin-receptor antagonist, prostacyclin analogue, phosphodiesterase type 5 inhibitor, or nitric oxide donor.
* Severe allergic reaction to iodine contrast
* Subjects receiving CYP3A4 and CYP2C9 inhibitors or inducers such as rifampin, ritonavir, fluconazole, amiodarone
* Not able to read or understand the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of pulmonary artery occlusion (Residual pulmonary vascular occlusion or RPVO) | 3 months
  To quantify RPVO we will use the Qanadli index (QI). The Qanadli index divides each pulmonary artery (right and left) into 10 segments. The presence of a thrombus in a segmental artery is scored with 1 point, a thrombus in the most proximal arterial level is scored with a value equal to the number of segmental arteries arising from that artery. The degree of obstruction score is obtained as follows: 0 when no thrombus, 1 is partially occlusive, and 2 is totally occlusive. The maximum possible index is 40. The percentage of obstruction is calculated using the following formula: % = QI Score /40 x 100. Percent of obstruction will be calculated at baseline and 3-month CT scan. The difference between 3 month-baseline percent of occlusion will be compared between Macitentan and placebo groups.

SECONDARY OUTCOMES:
The difference in levels of biomarkers of endothelial dysfunction and vascular remodeling | 3 months
  We will measure markers of endothelial dysfunction (CD31, CD41, CD62, CD144, CD54), change in diameter of brachial artery in millimeters from the flow mediated vasodilatation test (FMDba), FeNO levels in PPM and biomarkers of NO metabolism (ROS, ADMA, L-Arginine, Citrulline, NO and NOx) at baseline and at 3 months. We will compare the difference between 3-month -baseline values between the Macitentan and the placebo groups.
The difference in scores of functional capacity and severity of pulmonary hypertension | 6 months
  We will obtain questionnaires of quality of life (SF-36 and PEmb), a six-minute walking test, and the pulmonary pressure by echocardiogram, at baseline and 3-month visit. The difference between 3-month and baseline will be compared between the Macitentan and placebo groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No